CLINICAL TRIAL: NCT01278329
Title: Effect of Maternal Ante-natal Music Exposure on Neonatal Behavior Measured Using Brazelton Neonatal Behavioral Scale: A Randomized Open-label Study
Brief Title: Maternal Music Exposure During Pregnancy Influences Neonatal Behaviour
Acronym: PEXMUSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NSCB Medical College (Other)
Responsible Party: Maya Chansoria, NSCB Medical College, Jabalpur, MP, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEXMUSIC
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: Normal Healthy Term Appropriate-for-date Newborn
Keywords: Music; Foetal learning; Brazelton Neonatal Behavioral Assessment Scale

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music (Experimental): Mothers in the music group were provided a pre-recorded "Garbh Sanskar" audio cassette (Times Music Inc., Mumbai, India) with a running duration of approximately 50 minutes and a cassette player with headphones. They were asked to listen to the recorded music daily in the evening just before going to the bed with a minimum of ambient noise.
  Interventions: Other: "Garbh Sanskar" audio cassette (Times Music Inc., Mumbai, India)
- Control (No Intervention): Standard routine ante-natal care.

INTERVENTIONS:
Other: "Garbh Sanskar" audio cassette (Times Music Inc., Mumbai, India) — Approximate playing time = 50 minutes. Mothers advised to listen to it once every day.
  Arms: Music

SUMMARY:
Auditory stimulation during pregnancy has been found to influence foetal behaviour with a potential of being carried forward to neonatal period. This study evaluated the effect of ante-natal music exposure to primigravida healthy mothers on the behaviour of their term appropriate-for-date newborns. This was a single centre, randomized, open-label controlled trial. Primigravida mothers aged 19-29 years, free of chronic medical diseases or significant deafness, with singleton pregnancy, with a gestation of 20 weeks or less were randomized to listen to a pre-recorded music cassette for approximately 1 hour/day in addition to standard ante-natal care (intervention arm) or standard care only (control arm). Peri-natal factors with adverse effect on neonatal behaviour were deemed as protocol violations. The infants born to mothers exposed to music during pregnancy performed significantly better on 5 of the 7 BNBAS clusters. The maximal beneficial effect was seen with respect to orientation and habituation.

Conclusion:

Music exposure to mother during pregnancy significantly influences neonatal behaviour.

DETAILED DESCRIPTION:
Objective:

Auditory stimulation during pregnancy has been found to influence foetal behaviour with a potential of being carried forward to neonatal period. This study evaluated the effect of ante-natal music exposure to primigravida healthy mothers on the behaviour of their term appropriate-for-date newborns assessed using Brazelton Neonatal Behavioral Assessment Scale (BNBAS).

Methods:

This was a single centre, randomized, open-label controlled trial. Primigravida mothers aged 19-29 years, free of chronic medical diseases or significant deafness, with singleton pregnancy, with a gestation of 20 weeks or less were randomized to listen to a pre-recorded music cassette for approximately 1 hour/day in addition to standard ante-natal care (intervention arm) or standard care only (control arm). Peri-natal factors with adverse effect on neonatal behaviour were deemed as protocol violations. Outcome measure included scores on 7 clusters of BNBAS. Primary analysis was per protocol.

Results:

One hundred and 26 newborns in the music group and 134 in the control group were subjected to BNBAS assessment. The infants born to mothers exposed to music during pregnancy performed significantly better on 5 of the 7 BNBAS clusters. The maximal beneficial effect was seen with respect to orientation (ES 1.13, 95% CI 0.82-1.44, p<0.0001) and habituation (ES 1.05, 95% CI 0.53-1.57, p=0.0001).

Conclusion:

Music exposure to mother during pregnancy significantly influences neonatal behaviour.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive primigravida mothers of 19 to 29 years of age with singleton pregnancy attending the ante-natal clinic of the study institution first time, before 20 weeks of gestation were eligible for inclusion.

Exclusion Criteria:

* Mothers with significant co-existing medical diseases or severe to profound hearing loss were excluded

Ages: 19 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 339 (Actual)
Dates: Start 2003-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Performance on Brazelton Neonatal Behavioral Assessment Scale (BNBAS) | Day 2 or 3 of life
  Outcome measures consisted of the performance on Brazelton Neonatal Behavioral Assessment Scale (BNBAS). The BNBAS is a means of scoring interactive behaviour for term and stable preterm infants. The scale consists of 27 behavioural items, each scored on a 9-point scale, and 20 elicited responses, each scored on a 3-point scale. In most cases, the infant's score is based on the best performance, not an average performance.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Chansoria, MD, Study Director — NSCB Medical College
Locations (1):
- NSCB Medical College, Jabalpur, Madhya Pradesh, India

REFERENCES:
- [Derived] Arya R, Chansoria M, Konanki R, Tiwari DK. Maternal Music Exposure during Pregnancy Influences Neonatal Behaviour: An Open-Label Randomized Controlled Trial. Int J Pediatr. 2012;2012:901812. doi: 10.1155/2012/901812. Epub 2012 Feb 14. PMID 22518187